CLINICAL TRIAL: NCT05799625
Title: An Interactive Smartphone Application to Motivate Smokers to Quit
Acronym: StepOne
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20220696-01H
Record Dates: First submitted 2023-03-06; First posted 2023-04-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation; Smoking Behaviors
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Eligible smokers randomized to usual care will receive an educational brochure for the University of Ottawa Heart Institute's Ottawa Model for Smoking Cessation (OMSC) Community Program. The brochure will include information about the OMSC Community Program and how to register for it to receive assistance to quit smoking.
- Intervention (Experimental): Eligible smokers randomized to the intervention group will be asked to download the StepOne smartphone application onto their smartphone via the Apple Store or Google Play Store. They will be provided with a unique ID and unique code, which will enable them to log into the StepOne smartphone application to begin the 14-day program. Users will interact with the application in the morning and evening; the exact time of the engagement is selected by the participant and ideally at a time that maximizes the likelihood of engaging with the activity. The application incorporates interactive educational material, daily reminders, gamification, and models of habit formation to engage users. As with any other smartphone application, users can turn off notifications if they choose to do so. New content and activities will be shared daily.
  Interventions: Behavioral: StepOne Smartphone Application

INTERVENTIONS:
Behavioral: StepOne Smartphone Application — This smartphone application provides a 14-day program that delivers the core components of smoking cessation (i.e., counseling, education) and takes advantage of pandemic-accelerated acceptance of virtual care, videoconferencing, remote monitoring, and social networking. The program seeks to move participants from the pre-action stage (not interested in quitting) to the action stage (intention to quit) and incorporates daily reminders, gamification, and models of habit formation to engage users.
  Arms: Intervention

SUMMARY:
Prospective, randomized, single-blinded, blinded-endpoint trial to determine the impact of a smartphone application-based program to motivate smokers to increase readiness to quit, make quit attempts, and quit smoking.

DETAILED DESCRIPTION:
Prospective, randomized, single-blinded, blinded-endpoint trial to determine the impact of a smartphone application-based program to motivate smokers to increase readiness to quit, make quit attempts, and quit smoking. The intervention has been designed based by a team of scientist, taking principles of change behaviour into consideration. The application incorporates daily reminders, gamification, and models of habit formation to engage users. It will support participants to reflect on their smoking in a holistic manner through questions and activities.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Living in Ontario, Canada.
* Current smoker who indicates they are not interested in quitting within the next 30-days.
* Have access to and regularly use a smartphone with internet access.
* Read, write, speaks English or French.
* Available and willing to participate in follow-up assessments over the next 6 months.
* Able to provide consent.

Exclusion Criteria:

* Planning on quitting smoking within the next 30-days.
* Cognitively impaired or experiencing acute psychiatric illness that would alter their ability to participate.
* Institutionalized at a retirement home, nursing home or long-term care facility.
* Has morbid illness which will prevent completion of 6-month follow-up (e.g., receiving palliative care).
* Participating in another smoking cessation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported readiness to quit | Day 14
  Collected via survey
Self-reported readiness to quit | Day 45
  Collected via survey
Self-reported readiness to quit | Day 195
  Collected via survey
Having made a quit attempt | Day 14
  Collected via survey
Having made a quit attempt | Day 45
  Collected via survey
Having made a quit attempt | Day 195
  Collected via survey
Rate of smoking cessation | Day 45 for participants who report smoking cessation
  Biochemically verified using an expired carbon monoxide (CO) test
Rate of smoking cessation | Day 195 for participants who report smoking cessation
  Biochemically verified using an expired carbon monoxide (CO) test

SECONDARY OUTCOMES:
Number of participants that made a quit attempt | Day 14, 45, 195
  Collected via survey
Change in smoking | Day 14, 45, 195
  Collected via survey
Point prevalence abstinence | Day 14, 45, 195
  Collected via survey
Use of behavioural supports (e.g. counselling, quit lines) | Day 14, 45, 195
  Collected via survey
Use of cessation medication and/or e-cigarettes | Day 14, 45, 195
  Collected via survey
Satisfaction and perceived program barriers and facilitators will be assessed for patients in the intervention group | Day 14, 45, 195
  Collected via survey

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mir, MD, Principal Investigator — The University of Ottawa Heart Institute
Locations (1):
- The University of Ottawa Heart Institute, Ottawa, Ontario, Canada